CLINICAL TRIAL: NCT03241888
Title: Megestrol Acetate Plus LNG-IUS to Megestrol Acetate or LNG-IUS in Young Women With Endometrial Atypical Hyperplasia
Brief Title: Megestrol Acetate Plus LNG-IUS in Young Women With Endometrial Atypical Hyperplasia
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xiaojun Chen, Principal Investigator, Fudan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017-30-1
Record Dates: First submitted 2017-07-12; First posted 2017-08-08 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Atypical Endometrial Hyperplasia
Keywords: Levonorgestrel-releasing intrauterine system; megestrol acetate; Atypical Endometrial Hyperplasia
MeSH Terms: conditions — Endometrial Hyperplasia | interventions — Megestrol Acetate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MA (Active Comparator): Patients will receive megestrol acetate 160 mg by mouth daily for at least 3 months.Then every 3 months, an hysteroscope will be used to evaluate the endometrial condition, and the findings will be recorded.
  Interventions: Drug: Megestrol Acetate
- LNG-IUS (Active Comparator): Patients will receive LNG-IUS insertion for at least 3 months. Then every 3 months, an hysteroscope will be used to evaluate the endometrial condition, and the findings will be recorded.
  Interventions: Device: Levonorgestrel-releasing Intrauterine System(LNG-IUS)
- MA+LNG-IUS (Experimental): Patients will receive MA (160mg po qd) plus LNG-IUS insertion for at least 3 months. Then every 3 months, an hysteroscope will be used to evaluate the endometrial condition, and the findings will be recorded.
  Interventions: Drug: Megestrol Acetate; Device: Levonorgestrel-releasing Intrauterine System(LNG-IUS)

INTERVENTIONS:
Drug: Megestrol Acetate — At a dosage of 160 mg/day
  Other Names: Megace
  Arms: MA; MA+LNG-IUS
Device: Levonorgestrel-releasing Intrauterine System(LNG-IUS) — Active ingredient: levonorgestrel 52mg. It is a hormone-releasing T-shaped intrauterine system.
  Other Names: Mirena Intrauterine Device; Mirena
  Arms: LNG-IUS; MA+LNG-IUS

SUMMARY:
To see if megestrol acetate plus Levonorgestrel-releasing intrauterine system (LNG-IUS) will not be inferior to returning the endometrial tissue to a normal state than megestrol acetate or LNG-IUS alone in patients with endometrial atypical hyperplasia.

DETAILED DESCRIPTION:
After diagnosed of endometrial atypical hyperplasia (EAH) by hysteroscopy, patients will be enrolled. Age, waist circumstances, blood pressure, basic history of infertility, blood pressure, serum lipid level and side effects will be collected. Blood tests, including fasting blood glucose (FBG), postprandial blood glucose (PBG), fasting insulin (FINS), SHBG, sex hormone levels, blood lipids and anti-müllerian hormone(AMH) will be performed before treatment to evacuate their metabolic conditions.

Patients are randomized to 1 of 3 treatment groups. Patients will receive MA (megestrol acetate) 160 mg by mouth daily for at least 3 months on Arm I. Patients will receive LNG-IUS insertion on Arm II and MA 160 mg plus LNG-IUS insertion on Arm III. Then an hysteroscope will be used to evaluate the endometrial condition every 3 months, and the findings will be recorded. For patients with EAH, complete response (CR) is defined as the reversion of endometrial atypical hyperplasia to proliferative or secretory endometrium; partial response (PR) is defined as regression to simple or complex hyperplasia without atypia; no response (NR) is defined as the persistence of the disease; and progressive disease (PD) is defined as the appearance of endometrial cancer in patients. Continuous therapies will be needed in PR, NR or PD.

After completion of study treatment, 2 months of maintenance treatment will be recommended for patients with CR, and participants will be followed up for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Primarily have a confirmed diagnosis of endometrial atypical hyperplasia based upon hysteroscopy
* Have a desire for remaining reproductive function or uterus
* Need to be able to undergo correlative treatment and follow-up

Exclusion Criteria:

* Acute liver disease or liver tumor (benign or malignant) or renal dysfunction
* Pregnancy or suspicion of pregnancy
* Have a history of EAH and have disease relapse during Merina insertion
* Under treatment of high-dose progestin therapy more than 3 months in recent 6 months
* Congenital or acquired uterine anomaly including fibroids if they distort the uterine cavity
* Confirmed diagnosis of malignant tumor in genital system
* Acute severe disease such as stroke or heart infarction or a history of thrombosis disease
* Hypersensitivity or contradiction to any component of this product
* Ask for removal of the uterus or other conservative treatment
* Smoker(>15 cigarettes a day)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2017-07-04 (Actual); Primary Completion 2020-06-18 (Actual); Study Completion 2020-06-18 (Actual)

PRIMARY OUTCOMES:
Pathological response rate | From date of randomization until the date of CR or date of hysterectomy, whichever came first, assessed up to 12 months
  the proportion of histologic regression from endometrial atypical hyperplasia to benign endometrium
Pathological response time | From date of randomization until the date of CR or date of hysterectomy, whichever came first, assessed up to 12 months
  time of histologic regression from endometrial atypical hyperplasia to benign endometrium

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | up to 2 years after the treatment for each patient
  Common side effects from these drugs include weight gain, vaginal spotting and descent of sexuality. Severe side effects include thrombus and diseases related. The investigators will record any mental or body symptoms and evaluate the correlation.
Rate of relapse | up to 2 years after the treatment for each patient
  the proportion of experiencing recurrence after regression
Rate of pregnancy | up to 2 years after the treatment for each patient
  the proportion of getting pregnancy after regression
Compliance | up to 2 years after the treatment for each patient
  The investigators designed a questionnaire to evaluate the compliance through treatment as side effects of oral megestrol acetate may be more common than LNG-IUS. Self Efficacy, physical activity and social support will be scored (1 to 5) and compared among each arm.

OTHER OUTCOMES:
Economic consequences through study completion | From date of randomization until the date of CR or date of hysterectomy, whichever came first, assessed up to 12 months
  The investigators will evaluate whether the combination could shorten the therapeutic period, so that bring economic benefits.

CONTACTS AND LOCATIONS:
Locations (1):
- Obstetrics and Gynecology Hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Study data are available after a request email with indications.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The data are available since the publication of the study paper.
Access Criteria: The data can be accessed through email request.

REFERENCES:
- [Background] Gressel GM, Parkash V, Pal L. Management options and fertility-preserving therapy for premenopausal endometrial hyperplasia and early-stage endometrial cancer. Int J Gynaecol Obstet. 2015 Dec;131(3):234-9. doi: 10.1016/j.ijgo.2015.06.031. Epub 2015 Sep 8. PMID 26384790
- [Background] Park JY, Kim DY, Kim JH, Kim YM, Kim KR, Kim YT, Seong SJ, Kim TJ, Kim JW, Kim SM, Bae DS, Nam JH. Long-term oncologic outcomes after fertility-sparing management using oral progestin for young women with endometrial cancer (KGOG 2002). Eur J Cancer. 2013 Mar;49(4):868-74. doi: 10.1016/j.ejca.2012.09.017. Epub 2012 Oct 13. PMID 23072814
- [Background] Orbo A, Vereide A, Arnes M, Pettersen I, Straume B. Levonorgestrel-impregnated intrauterine device as treatment for endometrial hyperplasia: a national multicentre randomised trial. BJOG. 2014 Mar;121(4):477-86. doi: 10.1111/1471-0528.12499. Epub 2013 Nov 28. PMID 24286192
- [Background] Wildemeersch D, Janssens D, Pylyser K, De Wever N, Verbeeck G, Dhont M, Tjalma W. Management of patients with non-atypical and atypical endometrial hyperplasia with a levonorgestrel-releasing intrauterine system: long-term follow-up. Maturitas. 2007 Jun 20;57(2):210-3. doi: 10.1016/j.maturitas.2006.12.004. Epub 2007 Jan 31. PMID 17270370
- [Background] Montz FJ, Bristow RE, Bovicelli A, Tomacruz R, Kurman RJ. Intrauterine progesterone treatment of early endometrial cancer. Am J Obstet Gynecol. 2002 Apr;186(4):651-7. doi: 10.1067/mob.2002.122130. PMID 11967486
- [Background] Chen M, Jin Y, Li Y, Bi Y, Shan Y, Pan L. Oncologic and reproductive outcomes after fertility-sparing management with oral progestin for women with complex endometrial hyperplasia and endometrial cancer. Int J Gynaecol Obstet. 2016 Jan;132(1):34-8. doi: 10.1016/j.ijgo.2015.06.046. Epub 2015 Oct 1. PMID 26493012
- [Derived] Xu Z, Yang B, Shan W, Liao J, Shao W, Wu P, Zhou S, Ning C, Luo X, Zhu Q, Zhang H, Ma F, Guan J, Chen X. Comparison of the effect of levonorgestrel-intrauterine system with or without oral megestrol acetate on fertility-preserving treatment in patients with atypical endometrial hyperplasia: A prospective, open-label, randomized controlled phase II study. Gynecol Oncol. 2023 Jul;174:133-141. doi: 10.1016/j.ygyno.2023.05.001. Epub 2023 May 12. PMID 37182434
- [Derived] Mittermeier T, Farrant C, Wise MR. Levonorgestrel-releasing intrauterine system for endometrial hyperplasia. Cochrane Database Syst Rev. 2020 Sep 6;9(9):CD012658. doi: 10.1002/14651858.CD012658.pub2. PMID 32909630